CLINICAL TRIAL: NCT06574880
Title: STARLiT: STereotActic Body Radiotherapy and 177Lutetium PSMA in Locally Advanced Prostate Cancer: A Phase I/II Trial
Brief Title: STereotActic Body Radiotherapy and 177Lutetium PSMA in Locally Advanced Prostate Cancer
Acronym: STARLiT
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Angela Y. Jia, MD PhD (Other)
Responsible Party: Sponsor-Investigator, Angela Y. Jia, MD PhD, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE7824
Record Dates: First submitted 2024-08-26; First posted 2024-08-28 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Malignant Neoplasm of Prostate; Locally Advanced Prostate Cancer
Keywords: Prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Pluvicto

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lu-PSMA-617 + SBRT (Experimental): * Lu-PSMA-617: 7.4GBq intravenous infusion once with cycle 1, followed by 7.4GBq cycle 2 that is delivered 6 weeks after SBRT , and potentially 7.4GBq cycle #3 delivered 6 weeks after cycle #2 pending dose escalation
  * Radiation therapy: 5 fractions to prostate and elective nodal irradiation, SBRT, delivered 6 weeks after cycle 1 of 177Lu-PSMA-617
  Interventions: Drug: Lu-PSMA-617; Radiation: 5-fraction Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Drug: Lu-PSMA-617 — Lu-PSMA will be administered at a fixed dose of 7.4GBq per cycle, on a dose escalation schedule:
  * Level 0: Lu-PSMA-617 for 1 cycle, followed 6 weeks later by SBRT.
  * Level 1 (Starting Dose Level): Lu-PSMA-617 for 1 cycle, followed 6 weeks later by SBRT, followed 6 weeks later by cycle 2.
  * Level 2: Lu-PSMA-617 for 1 cycle, followed 6 weeks later by SBRT, followed 6 weeks later by cycle 2, followed 6 weeks later by cycle 3.
  Other Names: Pluvicto
Radiation: 5-fraction Stereotactic Body Radiation Therapy (SBRT) — Prostate and nodal SBRT will begin at the completion of cycle 1 (6 weeks after the first Lu-PSMA-617 infusion, ± 4 weeks).
  Other Names: SBRT

SUMMARY:
The goal of this clinical trial is to is to investigate if it is possible to lower the chance of cancer reoccurrence and also preserve quality of life by using the drug Pluvicto instead of androgen-deprivation therapy to the usual radiation therapy for advanced local prostate cancer.

Participants will receive one dose of Pluvicto, followed by radiation about 6 weeks later. Radiation therapy will be completed in 5 treatments over the period of 2 weeks. A second dose of Pluvicto will be given 6 weeks after radiation is complete. Some participants may also receive a third dose of Pluvicto, and this would be given 6 weeks after the second dose of Pluvicto.

DETAILED DESCRIPTION:
Prostate cancer is the most common cancer in men worldwide and second leading cause of cancer death in men. The most common treatment for prostate cancer is radiation therapy (RT) plus long-term androgen deprivation therapy (ADT) for 18-36 months with a consideration for the addition of abiraterone acetate.

With the introduction of abiraterone and other second generation androgen signaling inhibitors (ARSIs) there is great interest in shortening the duration of systemic therapy. This interest stems from the high toxicity rates of ADT and substantial impact on patient-reported quality of life (QoL). The use of ADT is associated with some adverse events. Therefore, the combination of adverse event risks and decrease in quality of life associated with castration have resulted in decreased compliance to long term ADT and even ARSIs, where approximately 50% of patients with locally advanced disease either decline any ADT or stop treatment early. The goal of this clinical trial is to is to investigate if it is possible to lower the chance of cancer reoccurrence and also preserve quality of life by using the drug Pluvicto instead of androgen-deprivation therapy to the usual radiation therapy for advanced local prostate cancer.

This clinical trial will evaluate the safety of using Lu-PSMA-617 with SBRT to the prostate and pelvic lymph nodes, and to determine whether Lu-PSMA-617 can replace androgen deprivation therapy (ADT) to improve oncologic outcomes by use of cytotoxic agents, avoid ADT related side effects, and improve compliance for participants to receive systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be ≥ 18 years of age.
* ECOG performance status ≤ 1
* Histologic confirmation of prostate adenocarcinoma of the prostate
* PSMA avid disease on PSMA PET/CT, where the tumor in the prostate has SUVmax ≥ 10.

  * PSMA PET/CT must be obtained within 4 months.
* Need ≥ 1 criteria:

  * Node positive disease on PSMA PET/CT or conventional imaging, as defined by having any of the following:

    * Pelvic nodal disease (cN1) as defined by LN stations that commence at the bifurcation of the common iliac vessels
    * Regional nodal disease (M1a) as defined by LN stations that commence at the bifurcation of the aorta and bifurcation of the proximal inferior vena cava to the common iliac veins.
  * In the absence of nodal metastasis, must have ≥ 2 of the following

    * i. cT3a or cT3b by conventional imaging (MRI) or PSMA PET/CT
    * ii. Grade group ≥ 4
    * iii. PSA ≥ 40 ng/mL
* Adequate organ and marrow function to receive treatment:

  * Hemoglobin > 10 g/dL
  * White blood cell (WBC) > 3000 / mL
  * Absolute neutrophil count ≥ 1,500 / mcL
  * Platelets ≥ 100,000 / mcL
  * Creatinine ≤ 1.5x ULN
  * Estimated glomerular filtration rate (eGFR)* > 50 mL/min
  * Total bilirubin** < 2× ULN
  * Albumin > 3 g/dL
  * Aspartate aminotransferase (AST) < 3× ULN

    * *based upon Chronic Kidney Disease- Epidemiology Collaboration (CKD-EPI) equation. Participants with estimated GFR between 50 - 60 mL/min will require a 99mTc-TPA GFR test and only participants with non-obstructive pathology will be included in the study.
    * ** Total bilirubin ≤ 2x ULN (except for participants with known Gilbert's Syndrome ≤ 3x ULN is permitted)
* International Prostate Symptoms Score (IPSS) ≤ 15.
* Medically fit for treatment and agreeable to follow-up.
* Ability to understand and the willingness to sign a written informed consent.
* Participants with partners of childbearing potential, agreement to use barrier contraceptive method (condom) and to continue its use for 14 weeks from receiving the last dose of Lu-PSMA-617. Participants must also not donate sperm for 14 weeks from receiving the last dose of Lu-PSMA-617.

Exclusion Criteria:

* Clinical or radiographic evidence of distant metastatic disease (M1a above aortic bifurcation, M1b, or M1c) by any imaging. Participants are allowed to M1a nodal disease that is below the aortic bifurcation. Negative PSMA PET/CT is an acceptable substitute to conventional staging.
* Prostate gland size >90 cc measured by CT, ultrasound, or MRI
* Prior head and neck radiation therapy.
* Prior treatment for prostate cancer (incudes chemotherapy, radiation therapy, or anti-androgen therapy).
* Prohibited within 30 days prior to administration to study treatment: spironolactone and other investigational drug therapies.
* Prohibited 3 months before participant registration and during administration of study treatment: oral ketoconazole, , estrogens, and radiopharmaceuticals.
* History of prior pelvic radiation therapy.
* Enrollment concurrently in another investigational drug study within 6 months of registration.
* History of another active malignancy within the previous 3 years except for adequately treated skin cancer or superficial bladder cancer.
* History of prior myelodysplastic syndrome or acute leukemia.
* History of or active Crohn's disease or ulcerative colitis.
* Contraindication to or inability to tolerate PSMA/PET.
* Any condition that in the opinion of the investigator would preclude participation in this study.
* Inability to adhere to radiation safety measures in hospital or at home
* Prior treatment with radionuclide therapies, 177Lu-PSMA-617 or other
* Reduced salivary gland function with baseline CTCAE Gr > 1 dry mouth will be excluded.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Phase I: Maximum tolerated dose (MTD) of Lu-PSMA-617 | 4 weeks after final dose of treatment (treatment expected to last up to six months)
  The Phase I goal is to determine the maximally tolerated dose (MTD) of Lu-PSMA-617 when administered with prostate SBRT treatment. The MTD will be captured by analyzing the incidence of dose limiting toxicities occurring within the four weeks after the last dose of treatment.
Phase II: Androgen deprivation therapy (ADT)-free survival | 3 years post treatment
  The Phase II goal is to determine the 3-year rate of ADT-free survival.

SECONDARY OUTCOMES:
PSA Progression Free Survival | 2 years post treatment
  PSA progression-free survival will be analyzed at 24 months post last dose of treatment.
Overall Survival (OS) | 5 years post treatment
  Overall Survival (OS) is defined as the time from Day 1 until death due to any cause. For subjects who do not die, time to death will be censored at the time of last contact.
Prostate Cancer-specific Survival (PCSM) | 5 years post treatment
  Prostate cancer specific mortality (PCSM) is defined the time from Day 1 to death directly attributable to prostate cancer, death from treatment complications, or death from unknown causes in participants with active prostate cancer or previously documented clinical or biochemical relapse.
Cumulative incidence of distant metastases | 5 years post treatment
  Distant metastases (DM) is defined as the time from Day 1 until development of distant metastases on CT, MRI, bone scan or PSMA PET, or death from prostate cancer.
Time to any salvage therapy | 5 years post treatment
  The time to any salvage therapy, or Time-to-next-intervention (TTNI), is defined as is defined as the time from Day 1 to the time of initiation of any additional (i.e., outside of planned protocol treatment) cancer-directed therapy, including but not limited to androgen deprivation, other systemic prostate cancer therapeutics, palliative radiotherapy, or surgical intervention specifically addressing complications of metastases. In the absence of a defining event, TTNI will be censored at the date of last visit documenting absence of interventions.
Change in Quality of life score as measured by EPIC-26 | Baseline to 5 years post treatment
  EPIC-26 is a short form version of the full Expanded Prostate Cancer Index Composite (EPIC). This version contains 26 items and the same 5 domains as the full version of EPIC: urinary incontinence, urinary irritative/obstructive, bowel, sexual, and hormonal. Response options for each EPIC item for a Likert scale, and multi-item scare scores are transported linearly to a 0-100 scale with higher scores representing better QoL. The time frame asked in the question relates to symptoms experienced within the prior 4 weeks.
Change in Quality of life score as measured by XeQoLS | Baseline to 5 years post treatment
  Xerostomia-related Quality of Life Questionnaire (XeQoLS) is a questionnaire used to measure how dry mouth and salivary dysfunction affect participants' quality of life (QoL). This questionnaire consists of 15 questions across four major domains: physical functioning, personal/psychological functioning, social functioning, and pain/discomfort issues. The XeQoLS is a self-administered tool, and participants are asked to rate each symptom on a 5-point Likert scale from 0 to 4, with higher scores indicating increased xerostomia burden. An average of scores in each domain is calculated, and the average score ranges from 0 to 4. A total score is calculated as an average of the scores from each of the domain.
Change in Quality of life score as measured by FACT-RNT | Baseline to 5 years post treatment
  FACT-RNT is a patient-reported outcomes (PRO) measure for PCa participants receiving radionuclide therapy. It has not yet been validated in a prospective manner. It consists of 15 questions on a 5-point Likert scale, in a recall period of the past 7 days. Each item score is added, and the sum is linearly transformed to produce the final summary score ranging from 0 to 100, with higher scores representing better QoL.
Time-to-castration-resistant prostate cancer | 5 years post treatment
  To determine the average time-to-castration-resistant prostate cancer.
Rate of participants with post treatment PSA in goal range | 12 weeks post treatment
  Rate of obtaining a post-treatment PSA of ≤ 0.5 ng/mL following treatment with 177Lu-PSMA-617 and prostate and nodal SBRT.
Incidence of acute toxicity | 5 years post treatment
  The goal is to describe acute toxicity following treatment with Lu-PSMA-617 and prostate and nodal SBRT.
Incidence of late toxicity | 5 years post treatment
  The goal is to describe late treatment toxicity following treatment with Lu-PSMA-617 and prostate and nodal SBRT.
Biochemical recurrence (BCR) | 5 years post treatment
  To determine the rate of biochemical recurrence (BCR), defined as PSA nadir + 2 ng/mL.
Proportion of participants with PSA50-RR | 12 weeks post treatment
  The proportion of participants with PSA50-RR at 12 weeks post all treatment will be summarized with 95% confidence interval (CI), where PSA50-RR is defined as the proportion of men with a PSA reduction of at least 50% at 6 weeks after the last 177Lu-PSMA-617 treatment, compared with baseline PSA prior to 177Lu-PSMA-617 treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Y Jia, MD, PhD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center; Daniel E Spratt, MD, Study Chair — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlies publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Compiled and analyzed participant data will be published upon study completion. Publisher may request Protocol and Statistical Analysis Plan.
Access Criteria: To be shared with investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose.